CLINICAL TRIAL: NCT07207629
Title: Evaluation of Transthoracic Echocardiography Parameters and Their Changes in Blood Donor Volunteers
Acronym: EDoS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: GIRCI SOHO (Other); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NIMAO/2024-2/FC-01
Record Dates: First submitted 2025-02-10; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Hemorrhage; Trauma; Shock Hypovolemic
Keywords: hemorrhagic shock; echocardiography; velocity time integral
MeSH Terms: conditions — Hemorrhage; Wounds and Injuries; Shock; Shock, Hemorrhagic

STUDY DESIGN:
Intervention Model Description: Healthy volunteer experiencing blood depletion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental)
  Interventions: Diagnostic Test: Transthoracic Echocardiography measurements

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiography measurements — TTE will be performed before, just after and 15 minutes after a blood donation, with measurement of aortic VTI, E wave, e' wave, A wave and left ventricle global longitudinal strain

SUMMARY:
This study investigates the impact of blood donation on transthoracic echocardiography (TTE) parameters in healthy volunteers, aiming to enhance the understanding of hemodynamic changes associated with mild blood loss and assess non-invasive monitoring techniques for early hemorrhage detection. Conducted as a prospective, interventional study with minimal risk, this research is designed to simulate a controlled hemorrhage in a civilian setting, using voluntary blood donation as a model to study the physiological effects of blood loss of approximately 6 mL/kg.

Rationale and Background Hemorrhagic shock is a leading cause of preventable death in trauma patients, particularly among younger populations. The ability to rapidly detect and quantify blood loss is crucial in trauma management, as delayed or excessive resuscitation can lead to adverse outcomes, including multi-organ failure and coagulopathy. Traditional methods of monitoring blood volume and cardiac output, such as invasive catheterization or imaging techniques like CT scans, may not be feasible or practical in prehospital settings. TTE, particularly the measurement of the aortic time-velocity integral (TVI) using Doppler echocardiography, presents a non-invasive and potentially valuable tool for assessing cardiac output and detecting early hemodynamic changes due to blood loss.

Primary Objective The primary objective of this study is to evaluate whether the aortic TVI decreases by at least 10% following a controlled blood volume reduction during blood donation. This decrease in TVI could serve as a reliable marker of reduced cardiac output and might allow clinicians to detect mild to moderate blood loss in trauma patients non-invasively.

Secondary Objectives

The study also aims to examine additional echocardiographic parameters that may indicate changes in hemodynamic status following blood loss. Secondary objectives include measuring changes in:

Shock index (SI), calculated as the ratio of heart rate to systolic blood pressure, a parameter often associated with hypovolemia.

E-wave and e'-wave velocities, which reflect left ventricular filling pressures and diastolic function.

Ratios of E/e' and E/A, which are indicative of left ventricular diastolic function and filling pressures.

Global longitudinal strain of the left ventricle (GLS), which represents myocardial contractility.

Methods Healthy adult volunteers meeting eligibility criteria for blood donation are recruited from local blood donation centers. Participants undergo baseline TTE to measure the aortic TVI, E-wave, e'-wave, and other relevant parameters before donation. Following a blood donation procedure of approximately 450 mL (representing a 6 mL/kg blood loss for the average volunteer), TTE is repeated immediately after donation and then 15 minutes post-donation to capture any transient changes in cardiac output and ventricular function. Volunteers receive structured hydration and are observed for any adverse events.

Outcome Measures The primary outcome measure is a decrease of at least 10% in aortic TVI from baseline immediately following blood donation, which would confirm the sensitivity of TTE to detect mild hypovolemia. Secondary outcome measures include changes in the shock index, variations in Doppler-derived E and e' waves, and the E/e' and E/A ratios, assessed immediately and 15 minutes post-donation. The study will also monitor the global longitudinal strain (GLS) as an additional measure of left ventricular performance.

Statistical Analysis The required sample size was calculated to detect a 10% decrease in TVI with 90% power at a 5% significance level, resulting in a target enrollment of 66 participants. Descriptive statistics will be used for continuous variables, expressed as mean ± standard deviation or median and interquartile range as appropriate. Paired t-tests or Wilcoxon signed-rank tests will assess changes in parameters before and after blood donation. Each participant's response will be classified as positive if a decrease of at least 10% in TVI is observed, or negative if the decrease is below this threshold.

Potential Impact If successful, this study could validate the use of TTE-derived parameters, such as aortic TVI and shock index, as non-invasive markers for early detection of blood loss in trauma patients. By providing real-time insight into hemodynamic changes, this approach could improve decision-making in prehospital and emergency settings, allowing clinicians to tailor resuscitation strategies based on the actual volume of blood loss. This could reduce the risks associated with both under-resuscitation and over-resuscitation, ultimately improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult volunteers eligible for blood donation according to French Blood Establishment (EFS) standards.

Age between 18 and 40 years. Participants who have provided written, informed consent. Affiliated with or a beneficiary of a social security system.

Exclusion Criteria:

Obesity (BMI > 30 kg/m²) or underweight (BMI < 18 kg/m²). Body weight over 96 kg. History of valvular heart disease, ischemic heart disease, or congestive heart failure.

Known allergy to ultrasound gel. Current medications that could affect hemodynamic response to blood loss (e.g., antihypertensives, antiepileptics, NSAIDs).

Participation in other human research studies defined as Category 1. Subjects under legal protection, including guardianship or curatorship. Pregnant, lactating, or breastfeeding women. Conditions that contraindicate blood donation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
aortic VTI variation | At two time points: prior to blood donation (baseline) and at completion of donation (at catheter withdrawal) - at day 0, 15 minutes after baseline
  measured by apical 5 cavity TTE

SECONDARY OUTCOMES:
Shock index variation | At three time points: prior to blood donation (baseline), at completion of donation (at catheter withdrawal) at day 0, 15 minutes after baseline ; and 15 minutes after blood donation (at day 0, 30 minutes after baseline)
  heart rate divided per systolic blood pressure
E wave variation | At three time points: prior to blood donation (baseline) , at completion of donation (at catheter withdrawal) at day 0, 15 minutes after baseline ; and 15 minutes after blood donation at day 0, 30 minutes after baseline
  measured on 4 cavity apical TTE
e' wave variation | At three time points: prior to blood donation (baseline), at completion of donation (at catheter withdrawal) at day 0, 15 minutes after baseline and 15 minutes after blood donation at day 0, 30 minutes after baseline
  measured on 4 cavity apical TTE
A wave variation | At three time points: prior to blood donation (baseline), at completion of donation (at catheter withdrawal) at day 0, 15 minutes after baseline and 15 minutes after blood donation at day 0, 30 minutes after baseline
  measured on 4 cavity apical TTE
E/A ratio variation | At three time points: prior to blood donation (baseline), at completion of donation (at catheter withdrawal) at day 0, 15 minutes after baseline and 15 minutes after blood donation at day 0, 30 minutes after baseline
  calculation of the ratio of E and A measures
E/e' ratio variation | At three time points: prior to blood donation (baseline), at completion of donation (at catheter withdrawal) at day 0, 15 minutes after baseline and 15 minutes after blood donation at day 0, 30 minutes after baseline
  calculation of the ratio of E and e' measures
Left ventricle global longitudinal strain variation | At three time points: prior to blood donation (baseline), at completion of donation (at catheter withdrawal) at day 0, 15 minutes after baseline and 15 minutes after blood donation at day 0, 30 minutes after baseline
aortic VTI variation persistance | at day 0, 15 minutes after baseline and 15 minutes after blood donation, at day 0, 30 minutes after baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Occitanie, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lamia B, Ochagavia A, Monnet X, Chemla D, Richard C, Teboul JL. Echocardiographic prediction of volume responsiveness in critically ill patients with spontaneously breathing activity. Intensive Care Med. 2007 Jul;33(7):1125-1132. doi: 10.1007/s00134-007-0646-7. Epub 2007 May 17. PMID 17508199